CLINICAL TRIAL: NCT07074288
Title: Obstructive Sleep Apnea Non-PAP Outcomes and Viable Alternatives (OSANOVA): Comparison of Mandibular Advancement Device and Hypoglossal Nerve Stimulation Outcomes
Brief Title: Obstructive Sleep Apnea Non-PAP Outcomes and Viable Alternatives
Acronym: OSANOVA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Jay F. Piccirillo, MD, Professor of Otolaryngology, Washington University School of Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202502149
Record Dates: First submitted 2025-06-25; First posted 2025-07-20 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Obstructive Sleep Apnea
Keywords: Otolaryngology; Mandibular Advancement Device therapy; Hypoglossal Nerve Stimulation therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Mandibular Advancement Device (MAD) therapy (Experimental): This arm includes patients who will receive treatment with a mandibular advancement device, which is an accepted therapy for moderate obstructive sleep apnea (OSA) patients following intolerance, refusal, or failure of positive airway pressure (PAP) therapy.
  Interventions: Device: MAD
- Hypoglossal Nerve Stimulation (HGNS) therapy (Active Comparator): This arm consists of patients who will receive hypoglossal nerve stimulation therapy, another accepted treatment option for moderate obstructive sleep apnea (OSA) patients following intolerance, refusal, or failure of positive airway pressure (PAP) therapy.
  Interventions: Device: HGNS

INTERVENTIONS:
Device: MAD — MAD intervention involves the use of a mandibular advancement device, which is designed to reposition the lower jaw and tongue to keep the airway open during sleep.
  Arms: Mandibular Advancement Device (MAD) therapy
Device: HGNS — HGNS intervention involves a surgical procedure to implant a device that stimulates the hypoglossal nerve to prevent airway collapse during sleep.
  Arms: Hypoglossal Nerve Stimulation (HGNS) therapy

SUMMARY:
OSANOVA is a non-randomized clinical trial which aims to compare outcomes of mandibular advancement device (MAD) and hypoglossal nerve stimulation (HGNS) therapies in moderate-to-severe OSA patients who fail, decline, or are intolerant to positive airway pressure (PAP) therapy (referred to as PAP-failing patients).

The primary aim of the study is to compare the outcomes between PAP-failing moderate-to-severe OSA patients receiving MAD and those receiving HGNS therapy. Primary Outcome measures include changes in Pittsburgh Sleep Quality Index (PSQI) scores.

Secondary aims will help us describe the outcomes between PAP-failing moderate-to-severe OSA patients receiving MAD and those receiving HGNS therapy. Secondary outcome measures include:

* adverse events,
* Epworth Sleepiness Scale (ESS),
* Symptoms of Nocturnal Obstruction and Related Events (SNORE-25),
* patient-reported satisfaction,
* CGI-Improvement,
* the rate of subjects re-selecting the treatment, and
* the rate of subjects recommending the treatment. and
* changes in sleep study metrics (i.e., AHI, ODI, mean arterial saturation, and Time<90%),

DETAILED DESCRIPTION:
The study will enroll and follow a cohort of PAP-failing patients receiving MAD therapy and a second cohort receiving HGNS therapy. Baseline and post-intervention patient-reported outcome measures (PROMs) and standard sleep study parameters to evaluate and compare treatment efficacy will be captured.

Both MAD and HGNS are accepted treatments for moderate OSA patients following PAP intolerance, refusal, or failure. Current decision-making is based heavily on patient preference rather than well-defined evidence-based recommendations. Choosing the right therapy is a crucial aspect of treatment for OSA, a chronic and lifelong condition.

ELIGIBILITY:
Inclusion Criteria:

* Must consent to being a part of the study
* Must be willing and able to physically present to the our office site on the Hospital campus whenever necessary over the course of the study
* Able to read, write, speak, and understand English
* Willing to complete study surveys over the course of the study.
* Must have a diagnosis for moderate to severe OSA (AHI ≥15) with indications for PAP therapy OSA is stratified into mild (5 ≤ AHI ≤ 15), moderate (15 < AHI ≤ 30), and severe (AHI>30)
* Must have declined PAP therapy (unwillingness to use), failed PAP therapy (AHI > 15 on PAP), or are inadherent to PAP therapy (not using PAP ≥4 hours/night for ≥5 nights per week, also defined as intolerance to PAP)
* Age ≥ 18 years
* BMI ≤ 40 kg/m²
* Central/Mixed apneas contribute < 25% of AHI (Predominantly Obstructive Sleep Apnea)
* Willing to complete pre-intervention and post-intervention sleep studies
* Planning to obtain MAD or HGNS as part of clinical care

Exclusion Criteria:

* AHI > 65

  o The guidelines for HGNS usage were originally approved for an AHI upper limit of 65. We will not enroll anyone in the study with an AHI greater than 65.
* Dental conditions such as temporomandibular joint disease, periodontal disease, dental disease, insufficient dentition (edentulism) to support appliance retention, and inadequate range of motion of the jaw. Similarly, patients undergoing dental realignment (e.g., braces or retaining device) are not suitable candidates.
* Chronic nasal obstruction
* Individuals without manual dexterity to place and remove the device such as those afflicted with severe arthritis, or neuromuscular disease that affects dexterity.
* Prior intolerance to MAD
* Rapid therapy required: patients in whom rapid initiation of treatment is desirable (e.g., patients with severe symptomatic OSA, sleepiness while driving) and they declined PAP without PAP failure. PAP therapy can be initiated quickly while MAD initiation requires incremental titration of the device over weeks to months to attain optimal efficacy.
* Severe or prolonged Oxygen desaturation: patients with severe oxyhemoglobin desaturation during sleep (e.g., nadir peripheral oxygen saturation [SpO2] <70 percent), caution is warranted as oral appliance therapy may not provide optimal improvement in oxygenation.
* Alcohol or illicit substance use at least daily
* Unstable psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | baseline(pre-treatment) and through study completion on average 8 weeks
  Pittsburgh Sleep Quality Index (PSQI) asks patients to reflect on their sleep experiences over the last month prior to assessment. The global PSQI score is calculated by summing all seven components scores (i.e., subjective sleep quality,sleep latency, sleep duration, habitual sleep efficiency,sleep disturbances, use of sleeping medication and daytime dysfunction). Each component is scored between 0 and 3, resulting in a total PSQI score ranging from 0 to 21. A higher score indicates poorer sleep quality, with a global sum greater than 5 signifying poor sleep quality.
  The change in PSQI is calculated as the difference in PSQI score post-treatment minus PSQI score pre-treatment.

SECONDARY OUTCOMES:
Clinical Global Impressions-Improvement (CGI-I) | through study completion on average 8 weeks
  CGI-I scale is a tool used to assess the change in a patient's condition following treatment. It is adapted from the Clinical Global Impression of Improvement scale and specifically measures improvement in obstructive sleep apnea (OSA). Patients are asked to evaluate their current condition compared to their status prior to receiving therapy. The response options for the CGI-I include categories such as:
  * Very much improved,
  * Somewhat improved,
  * Minimally improved,
  * No change,
  * Minimally worse,
  * Somewhat worse,
  * Very much worse.
  This scale helps quantify the perceived effectiveness of the treatment from the patient's perspective during follow-up assessments.
  Patients responding at least "minimally improved improvement" will be defined as responders to treatment.
Epworth Sleepiness Scale (ESS) scores. | baseline (pre-treatment) and through study completion on average 8 weeks
  The Epworth Sleepiness Scale (ESS) is a self-reported questionnaire that measures daytime sleepiness. It consists of eight scenarios in which respondents rate their likelihood of dozing off or falling asleep on a scale from 0 to 3, with higher scores indicating greater levels of daytime sleepiness. The total score can range from 0 to 24, with scores above 10 typically suggesting excessive daytime sleepiness.
  ESS score is calculated as the difference in ESS score post-treatment minus ESS score pre-treatment.
Symptoms of Nocturnal Obstruction and Related Events (SNORE-25) scores. | baseline (pre-treatment) and through study completion on average 8 weeks
  The SNORE-25 is a measure of sleep-disordered breathing-related health burden over the past two weeks. It is derived from a 7-item reduction of the OSA Patient-Oriented Severity Index (OSAPOSI). The SNORE-25 uses a magnitude scale ranging from 0 to 5 for each of its twenty-five items, resulting in a final score range of 0 to 125.
  A clinically meaningful difference is a 50% change (decrease) from pretreatment.
  The change in SNORE-25 is calculated as the difference in SNORE-25 score post-treatment minus SNORE-25 pre-treatment.
Measure of satisfaction with treatment | and through study completion on average 8 weeks
  Measure of satisfaction with treatment will capture global indication of satisfaction with the treatment.
  Response options are:
  * Very dissatisfied,
  * Mildly satisfied,
  * Neither satisfied or dissatisfied,
  * Mildly satisfied, , and
  * Very satisfied
The rate of subject re-selecting the treatment | and through study completion on average 8 weeks
  Response options are:
  * I would definitely select this treatment again,
  * I would likely select this treatment again,
  * I would likely not select this treatment again,
  * I would never select this treatment again.
  The rate of subjects responding "…definitely select this treatment again" and"…likely select this treatment again" will be compared between the two study group.
The rate of subjects recommending the treatment | and through study completion on average 8 weeks
  Response options are:
  * I would definitely recommend this treatment,
  * I would likely recommend this treatment,
  * I would likely not recommend this treatment,
  * I would never recommend this treatment,
  The rate of subjects responding "…definitely recommend this treatment" and "…likely recommend this treatment" will be compared between the two study groups.
Apnea-Hypopnea Index (AHI) | baseline (pre-treatment) and through study completion on average 8 weeks
  AHI is a measure of breathing interruptions during sleep. A higher AHI indicates more frequent breathing disruptions and more severe sleep apnea. A reduction in AHI indicates improved sleep apnea
Oxygen Desaturation Index (ODI) | baseline (pre-treatment) and through study completion on average 8 weeks
  ODI is a measure of oxygen desaturations during sleep. A reduction in ODI indicates improved sleep apnea.
Mean arterial saturation | baseline (pre-treatment) and through study completion on average 8 weeks
  Mean arterial saturation, which is a measure of peripheral artery oxygenation during sleep. An increase of mean arterial saturation indicates improved sleep apnea
Time <90% | baseline (pre-treatment) and through study completion on average 8 weeks
  This is a measure of the time spent below an oxygen saturation of 90% during sleep. A reduction in time < 90% indicates improved sleep apnea
Adverse events | throughout the entire study period on average 10 weeks
  Any undesirable experiences associated with the use of the intervention, which can include but are not limited to discomfort, pain, device-related issues, or other health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Jay F Piccirillo, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Basyuni S, Barabas M, Quinnell T. An update on mandibular advancement devices for the treatment of obstructive sleep apnoea hypopnoea syndrome. J Thorac Dis. 2018 Jan;10(Suppl 1):S48-S56. doi: 10.21037/jtd.2017.12.18. PMID 29445528
- [Background] Bentan MA, Nord R. Comprehensive Analysis of Adverse Events Associated With Hypoglossal Nerve Stimulators: Insights From the MAUDE Database. Otolaryngol Head Neck Surg. 2024 Nov;171(5):1580-1590. doi: 10.1002/ohn.883. Epub 2024 Jun 29. PMID 38943447
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cistulli PA. Oral appliances in the treatment of obstructive sleep apnea in adults. In: Collop N, Finlay G, eds. UpToDate. Waltham, MA: UpToDate Inc. https://www.uptodate.com/contents/oral-appliances-in-the-treatment-of-obstructive-sleep-apnea-in-adults. Topic 7678, Version 38.0. Accessed October 30, 2024.
- [Background] de Vries GE, Hoekema A, Vermeulen KM, Claessen JQPJ, Jacobs W, van der Maten J, van der Hoeven JH, Stegenga B, Kerstjens HAM, Wijkstra PJ. Clinical- and Cost-Effectiveness of a Mandibular Advancement Device Versus Continuous Positive Airway Pressure in Moderate Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Oct 15;15(10):1477-1485. doi: 10.5664/jcsm.7980. PMID 31596213
- [Background] El-Solh AA, Moitheennazima B, Akinnusi ME, Churder PM, Lafornara AM. Combined oral appliance and positive airway pressure therapy for obstructive sleep apnea: a pilot study. Sleep Breath. 2011 May;15(2):203-8. doi: 10.1007/s11325-010-0437-1. Epub 2010 Nov 10. PMID 21063793
- [Background] Epstein LJ, Kristo D, Strollo PJ Jr, Friedman N, Malhotra A, Patil SP, Ramar K, Rogers R, Schwab RJ, Weaver EM, Weinstein MD; Adult Obstructive Sleep Apnea Task Force of the American Academy of Sleep Medicine. Clinical guideline for the evaluation, management and long-term care of obstructive sleep apnea in adults. J Clin Sleep Med. 2009 Jun 15;5(3):263-76. PMID 19960649
- [Background] Francis CE, Quinnell T. Mandibular Advancement Devices for OSA: An Alternative to CPAP? Pulm Ther. 2021 Jun;7(1):25-36. doi: 10.1007/s41030-020-00137-2. Epub 2020 Nov 10. PMID 33170490
- [Background] Glos M, Penzel T, Schoebel C, Nitzsche GR, Zimmermann S, Rudolph C, Blau A, Baumann G, Jost-Brinkmann PG, Rautengarten S, Meier JC, Peroz I, Fietze I. Comparison of effects of OSA treatment by MAD and by CPAP on cardiac autonomic function during daytime. Sleep Breath. 2016 May;20(2):635-46. doi: 10.1007/s11325-015-1265-0. Epub 2015 Oct 13. PMID 26463420
- [Background] Gonzalez Castro S, Pozuelo Sánchez L, Jara Alonso I, Pérez Figuera A, Muriel García A, Carreño Alejandre A, Parra Jarque M, Delgado Vera-Pinto L, García Sánchez A,Cano Pumarega I, Mañas Baena E. [Title of the article]. Eur Respir J. 2023;62(suppl 67). doi:10.1183/13993003.congress-2023.PA3012.
- [Background] Gotsopoulos H, Chen C, Qian J, Cistulli PA. Oral appliance therapy improves symptoms in obstructive sleep apnea: a randomized, controlled trial. Am J Respir Crit Care Med. 2002 Sep 1;166(5):743-8. doi: 10.1164/rccm.200203-208OC. PMID 12204875
- [Background] Guimaraes MLR, Hermont AP, Guimaraes TM, Dal-Fabbro C, Bittencourt L, Chaves Junior CM. Severe obstructive sleep apnea treatment with mandibular advancement device: A case report. Sleep Sci. 2018 Mar-Apr;11(2):118-122. doi: 10.5935/1984-0063.20180022. PMID 30083300
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Background] Kent D, Stanley J, Aurora RN, Levine C, Gottlieb DJ, Spann MD, Torre CA, Green K, Harrod CG. Referral of adults with obstructive sleep apnea for surgical consultation: an American Academy of Sleep Medicine clinical practice guideline. J Clin Sleep Med. 2021 Dec 1;17(12):2499-2505. doi: 10.5664/jcsm.9592. PMID 34351848
- [Background] Kline LR. Clinical presentation and diagnosis of obstructive sleep apnea in adults. In: Collop N, Finlay G, eds. UpToDate. Waltham, MA: UpToDate Inc. https://www.uptodate.com/contents/clinical-presentation-and-diagnosis-of-obstructive-sleep-apnea-in-adults. Topic 7706, Version 66.0. Accessed October 30, 2024.
- [Background] Lee CH, Mo JH, Choi IJ, Lee HJ, Seo BS, Kim DY, Yun PY, Yoon IY, Won Lee H, Kim JW. The mandibular advancement device and patient selection in the treatment of obstructive sleep apnea. Arch Otolaryngol Head Neck Surg. 2009 May;135(5):439-44. doi: 10.1001/archoto.2009.31. PMID 19451462
- [Background] Longo UG, Berton A, De Salvatore S, Piergentili I, Casciani E, Faldetta A, De Marinis MG, Denaro V. Minimal Clinically Important Difference and Patient Acceptable Symptom State for the Pittsburgh Sleep Quality Index in Patients Who Underwent Rotator Cuff Tear Repair. Int J Environ Res Public Health. 2021 Aug 17;18(16):8666. doi: 10.3390/ijerph18168666. PMID 34444415
- [Background] Malhotra A, Kundel V. Obstructive sleep apnea: Overview of management in adults. In: Collop N, Finlay G, eds. UpToDate. Waltham, MA: UpToDate Inc. https://www.uptodate.com/contents/obstructive-sleep-apnea-overview-of-management-in-adults. Topic 7695, Version 108.0. Accessed October 30, 2024.
- [Background] Mehta A, Qian J, Petocz P, Darendeliler MA, Cistulli PA. A randomized, controlled study of a mandibular advancement splint for obstructive sleep apnea. Am J Respir Crit Care Med. 2001 May;163(6):1457-61. doi: 10.1164/ajrccm.163.6.2004213. PMID 11371418
- [Background] Patel S, Kon SSC, Nolan CM, Barker RE, Simonds AK, Morrell MJ, Man WD. The Epworth Sleepiness Scale: Minimum Clinically Important Difference in Obstructive Sleep Apnea. Am J Respir Crit Care Med. 2018 Apr 1;197(7):961-963. doi: 10.1164/rccm.201704-0672LE. No abstract available. PMID 28961021
- [Background] Piccirillo JF, Gates GA, White DL, Schectman KB. Obstructive sleep apnea treatment outcomes pilot study. Otolaryngol Head Neck Surg. 1998 Jun;118(6):833-44. doi: 10.1016/S0194-5998(98)70277-3. PMID 9627245
- [Background] Pietzsch JB, Liu S, Garner AM, Kezirian EJ, Strollo PJ. Long-Term Cost-Effectiveness of Upper Airway Stimulation for the Treatment of Obstructive Sleep Apnea: A Model-Based Projection Based on the STAR Trial. Sleep. 2015 May 1;38(5):735-44. doi: 10.5665/sleep.4666. PMID 25348126
- [Background] Quinnell TG, Bennett M, Jordan J, Clutterbuck-James AL, Davies MG, Smith IE, Oscroft N, Pittman MA, Cameron M, Chadwick R, Morrell MJ, Glover MJ, Fox-Rushby JA, Sharples LD. A crossover randomised controlled trial of oral mandibular advancement devices for obstructive sleep apnoea-hypopnoea (TOMADO). Thorax. 2014 Oct;69(10):938-45. doi: 10.1136/thoraxjnl-2014-205464. Epub 2014 Jul 17. PMID 25035126
- [Background] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920
- [Background] Randerath W, Verbraecken J, de Raaff CAL, Hedner J, Herkenrath S, Hohenhorst W, Jakob T, Marrone O, Marklund M, McNicholas WT, Morgan RL, Pepin JL, Schiza S, Skoetz N, Smyth D, Steier J, Tonia T, Trzepizur W, van Mechelen PH, Wijkstra P. European Respiratory Society guideline on non-CPAP therapies for obstructive sleep apnoea. Eur Respir Rev. 2021 Nov 30;30(162):210200. doi: 10.1183/16000617.0200-2021. Print 2021 Dec 31. PMID 34853097
- [Background] Rotenberg BW, Murariu D, Pang KP. Trends in CPAP adherence over twenty years of data collection: a flattened curve. J Otolaryngol Head Neck Surg. 2016 Aug 19;45(1):43. doi: 10.1186/s40463-016-0156-0. PMID 27542595
- [Background] Stern J, Lee K, Kuhns D, Martinez-Kratz JF. Efficacy and Effectiveness of the ProSomnus(R) [IA] Sleep Device for the Treatment of Obstructive Sleep Apnea: EFFECTS Study. Cureus. 2021 Jun 2;13(6):e15391. doi: 10.7759/cureus.15391. eCollection 2021 Jun. PMID 34249542
- [Background] Strollo PJ Jr, Soose RJ, Maurer JT, de Vries N, Cornelius J, Froymovich O, Hanson RD, Padhya TA, Steward DL, Gillespie MB, Woodson BT, Van de Heyning PH, Goetting MG, Vanderveken OM, Feldman N, Knaack L, Strohl KP; STAR Trial Group. Upper-airway stimulation for obstructive sleep apnea. N Engl J Med. 2014 Jan 9;370(2):139-49. doi: 10.1056/NEJMoa1308659. PMID 24401051
- [Background] Suurna M. Hypoglossal nerve stimulation for adult patients with obstructive sleep apnea. In: Collop N, Finlay G, eds. UpToDate. Waltham, MA: UpToDate Inc. https://www.uptodate.com/contents/hypoglossal-nerve-stimulation-for-adult-patients-with-obstructive-sleep-apnea. Topic 135053, Version 12.0. Accessed October 30, 2024.
- [Background] Vanderveken OM, Beyers J, Op de Beeck S, Dieltjens M, Willemen M, Verbraecken JA, De Backer WA, Van de Heyning PH. Development of a Clinical Pathway and Technical Aspects of Upper Airway Stimulation Therapy for Obstructive Sleep Apnea. Front Neurosci. 2017 Sep 21;11:523. doi: 10.3389/fnins.2017.00523. eCollection 2017. PMID 28983236
- [Background] Vecchierini MF, Attali V, Collet JM, d'Ortho MP, Goutorbe F, Kerbrat JB, Leger D, Lavergne F, Monaca C, Monteyrol PJ, Mullens E, Pigearias B, Martin F, Khemliche H, Lerousseau L, Meurice JC. Mandibular advancement device use in obstructive sleep apnea: ORCADES study 5-year follow-up data. J Clin Sleep Med. 2021 Aug 1;17(8):1695-1705. doi: 10.5664/jcsm.9308. PMID 34165074
- [Background] Verbraecken J, Dieltjens M, Op de Beeck S, Vroegop A, Braem M, Vanderveken O, Randerath W. Non-CPAP therapy for obstructive sleep apnoea. Breathe (Sheff). 2022 Sep;18(3):220164. doi: 10.1183/20734735.0164-2022. Epub 2022 Oct 11. PMID 36340820
- [Background] Weaver TE. Assessing and managing nonadherence with continuous positive airway pressure (CPAP) for adults with obstructive sleep apnea. In: Collop N, Finlay G, eds. UpToDate. Waltham, MA: UpToDate Inc. https://www.uptodate.com/contents/assessing-and-managing-nonadherence-with-continuous-positive-airway-pressure-cpap-for-adults-with-obstructive-sleep-apnea. Topic 7702, Version 50.0. Accessed October 30, 2024.
- [Background] Wojda M, Kostrzewa-Janicka J, Sliwinski P, Bielen P, Jurkowski P, Wojda R, Mierzwinska-Nastalska E. Mandibular Advancement Devices in Obstructive Sleep Apnea Patients Intolerant to Continuous Positive Airway Pressure Treatment. Adv Exp Med Biol. 2019;1150:35-42. doi: 10.1007/5584_2018_275. PMID 30255301
- [Background] Hughes CM, McCullough CA, Bradbury I, Boyde C, Hume D, Yuan J, Quinn F, McDonough SM. Acupuncture and reflexology for insomnia: a feasibility study. Acupunct Med. 2009 Dec;27(4):163-8. doi: 10.1136/aim.2009.000760. PMID 19942722